CLINICAL TRIAL: NCT07282015
Title: A Prospective Study to Describe the Real-world Treatment Outcomes in Canadian Patients With Moderate-to-severe Hidradenitis Suppurativa Treated With secukInumab (HS-RISE)
Brief Title: Real-world Secukinumab Outcomes in Canadian HS Patients
Acronym: HS-RISE
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MCA01
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; NIS; secukinumab; Phase IV
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Secukinumab: Patients with moderate-to-severe HS who are prescribed secukinumab in Canadian routine clinical practice

SUMMARY:
The HS-RISE study aims to assess real-world HS treatment outcomes and patterns, safety of secukinumab, and to describe the baseline characteristics of patients diagnosed with moderate-to- severe HS who are prescribed secukinumab in Canadian routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written, signed, and dated informed consent before any information is collected and any study-related activity is performed.
2. Adult patients at the time of informed consent signature.
3. Patients with the diagnosis of moderate-to-severe HS, as determined by the dermatologist.
4. Patients who have been newly prescribed secukinumab as part of routine clinical care according to the approved Canadian PM. The decision to prescribe secukinumab must be made prior to,and independent of, study participation. First treatment with secukinumab must occur no more than 7 days (≤7 days) prior to Baseline visit.
5. Patients who can understand written and spoken Canadian English or French.

Exclusion Criteria:

1. Any medical or psychological condition in the treating physician's opinion that may prevent the patient from study participation.
2. Patients who have any contraindications to treatment with secukinumab, as defined in the Canadian PM.
3. Patients who have had any prior exposure to secukinumab (i.e., >7 days prior to the baseline visit).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian patients diagnosed with moderate-to-severe HS and treated with secukinumab as per routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who experience a change in disease severity classification | Baseline, month 12
  Proportion of patients who experience a change in disease severity classification from baseline to 12 months, as determined by the International HS Severity Score System (IHS4).
  Determining IHS4 score requires counting nodules, abscesses and draining tunnels/sinus tracts. A score of 3 or less signifies mild HS, a score of 4 to 10 signifies moderate HS, and a score of 11 or higher signifies severe HS.

SECONDARY OUTCOMES:
Proportion of patients overall who experience a change in disease severity classification | Baseline, Month 3, Month 6
  Proportion of patients overall who experience a change in disease severity classification as determined by IHS4 from baseline at Months 3 and 6; additional subgroups analyses by ethnicity/race.
  Determining IHS4 score requires counting nodules, abscesses and draining tunnels/sinus tracts. A score of 3 or less signifies mild HS, a score of 4 to 10 signifies moderate HS, and a score of 11 or higher signifies severe HS.
Proportion of patients achieving a 55% reduction in International HS Severity Score System (IHS4-55) | Baseline, Month 3, Month 6, Month 12
  Proportion of patients achieving IHS4-55 at Months 3, 6, and 12; additional subgroups analyses by ethnicity/race.
  IHS4-55 is defined as at least a 55% reduction in their IHS4 from baseline.
Proportion of patients experiencing HS Clinical Response 50 (HiSCRO50) | Baseline, Month 3, Month 6, Month 12
  Proportion of patients achieving a 50% reduction from baseline in HS Clinical Response Score (HiSCR50) at Months 3, 6, and 12; additional subgroups analyses by ethnicity/race.
  HiSCR50 is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule (AN) count, with no increase from baseline in abscesses or draining fistulae count.
Mean reduction in abscess and inflammatory nodule count | Baseline, Month 3, Month 6, Month 12
  Mean reduction in abscess and inflammatory nodule count from baseline at Months 3, 6, and 12; additional subgroups analyses by ethnicity/race
Descriptive summaries of demographic and clinical variables | Baseline
  Descriptive summaries demographic and clinical variables
Proportion of patients receiving secukinumab up-titration from every 4 weeks (Q4W) to every 2 weeks (Q2W) | Month 3, Month 6, Month 12
  Proportion of patients receiving secukinumab up-titration from Q4W to Q2W at Months 3, 6, and 12; Subgroup analysis by ethnicity/race as well as time to biologic treatment initiation
Proportion of patients receiving secukinumab down-titration from every 2 weeks (Q2W) to every 4 weeks (Q4W) | Month 3, Month 6, Month 12
  Proportion of patients receiving secukinumab down-titration from Q2W to Q4W at Months 3, 6, and 12; Subgroup analysis by ethnicity/race as well as time to biologic treatment initiation
Time to secukinumab up- and down-titration | Month 3, Month 6, Month 12
  Time to secukinumab up- and down-titration
Proportion of patients experiencing adverse events post-secukinumab initiation | Up to 12 Months
  Proportion of patients experiencing adverse events post-secukinumab initiation
Proportion of patients experiencing serious adverse events post-secukinumab initiation | Up to 12 Months
  Proportion of patients experiencing serious adverse events post-secukinumab initiation
Type of adverse events and serious adverse events experienced by patients post-secukinumab initiation | Up to 12 Months
  Type of adverse events and serious adverse events experienced by patients post-secukinumab initiation
Proportion of patients who discontinued secukinumab due to adverse events | Up to 12 Months
  Proportion of patients who discontinued secukinumab due to adverse events
Proportion of patients receiving additional HS-related therapies | Month 3, Month 6, Month 12
  Proportion of patients receiving additional HS-related therapies at Months 3, 6, and 12; additional subgroup analysis by dosing, ethnicity/race and time to biologic initiation
Proportion of patients requiring unplanned surgeries | Month 3, Month 6, Month 12
  Proportion of patients requiring unplanned surgeries at Month 3, 6, and 12; additional subgroup analysis by dosing, ethnicity/race and time to biologic initiation
Proportion of patients discontinuing secukinumab treatment | Month 3, Month 6, Month 12
  Proportion of patients discontinuing secukinumab treatment at Months 3, 6, and 12; additional sugbroup analyses also done by ethnicity/race
Reason(s) for secukinumab discontinuation | Up to 12 Months
  Reason(s) for secukinumab discontinuation; additional subgroup analyses by ethnicity/race
Percentage of no-show appointments which were scheduled as per standard of care | Up to 12 Months
  Percentage of no-show appointments which were scheduled as per standard of care with participating dermatologist (including injections) and the corresponding reason(s); additional subgroup analyses by ethnicity/race

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Canada (7):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Richmond Hill, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No